## Statistical/Programming Plan for Cue Reward Trial Analysis

Protocol Version Date: 2022-12-16

1. Title: Medication Adherence Patterns in Rheumatic Diseases: A Behavioral Trial: Phase 2 trial results

## 2. Core research team

PI: Candace H Feldman; Co-PI: Niteesh Choudhry

3. Aim(s): To determine whether strategies that couple context cues and rewards improve adherence to medications

#### 4. Data source:

- a) REDCap data for 56 consented patients (20 = in Adaptive intervention; 18 = in Non-Adaptive Intervention; 18 = in Control) one dataset
- b) Pillsy pill bottle adherence data for 56 patients there are N= 352 daily 000\_Pillsy files spanning the length of the trial
- c) IRB: 2020P003826
- d) NIA (NIH) funded P30

## 5. Overall trial diagram:



### 6. Cohort Identification

### 6.1 Cohort Summary

There will be 1 cohort formed at the patient level.

Each patient should already be identified with the following in the REDCap dataset:

- e) Patient Study ID (i.e., Record id)
- f) Arm (arm) (0 = Control, 1 = Non-adaptive intervention, 2 = Adaptive intervention)

#### 6.2 Important steps for cohort formation

- 6.2.1 Eligible study entry dates/definitions and the corresponding variable names in REDCap.
  - a) **Screening date:** Date each patient was screened for eligibility for the study and began being contacted for enrollment. (mail date)
  - b) <u>Enrollment date:</u> Date each patient was enrolled and consented into the study. (date\_consent)
  - c) <u>Index date</u>: Each patient began receiving the intervention (either of the text messaging interventions or control). (start\_date)
  - d) Intervention Completion date: Index date (inclusive) to 12 weeks beginning on the index date (intervention date)
  - e) **Follow-up period**: Index date (inclusive) to 18 weeks beginning on the index date for primary adherence and secondary outcomes.

### 6.2.2 Specify <u>inclusion</u> criteria for cohort entry and define the index date

Patients are already identified by their study ID (56 patients altogether). The index date is the first day of intervention ("start\_date" in REDCap).

#### 7. Variables

### 7.1 Exposure-related variables:

**Patient-level cohort:** Within this cohort, please measure and provide the following variables at the patient level:

- a) Using the REDCap file:
  - Patient demographics:
    - Age (age\_years, age), numeric. Please also calculate using dob and start\_date
    - Sex (sex)
      - 0 = Not listed
      - 1 = Female
      - 2 = Male
    - Sex if Sex is not listed (sex\_other)
    - Race/ethnicity (self reported)
      - 1 = White
      - 2 = Black or African American
      - 3 = American Indian/ Alaska Native
      - 4 = Asian
      - 5 = Native Hawaiian or Other Pacific Islander
      - 6 = Hispanic/Latinx
    - Education level (education):
      - 1 = Less than high school diploma
      - 2 = High school diploma
      - 3 = Some college
      - 4 = College degree
      - 5 = Graduate degree
    - Marital status (marital)
      - 1 = Married
      - 2 = Living with partner/ Domestic partnership
      - 3 = Widowed
      - 4 = Divorced/ Separated
      - 5 = Never married/ Single
    - Employment Status (employment)
      - 1 = Employed
      - 2 = Job seeking

- 3 = Not job seeking
- 4 = Retired
- 5 = Disabled
- Income (self-reported) (income)
  - 1 = Less than \$20,000
  - 2 = \$20,000 to \$34,999
  - 3 = \$35,000 to \$49,999
  - 4 = \$50,000 to \$74,999
  - 5 = \$75,000 to \$99,999
  - 6 = Over \$100,000
  - 7 = Prefer not to say
- o Number of self-reported medications on a daily basis (num meds daily)
- Number of self-reported medications on a weekly basis (num\_meds\_weekly)
- Recruitment method (rec type)
  - 1 = PCP
  - 2 = Rheumatology
- Baseline Uric acid (ua\_baseline) used for the study, numeric
- Baseline Uric acid date (ua baseline date)
- Baseline Uric acid stratum (ua stratum)
  - 1 = 6-8 mg/dl
  - 2 = >8 mg/dl
- O Arm (arm):
  - 0 = Control,
  - 1 = Non-adaptive intervention,
  - 2 = Adaptive intervention
- Number of prescribed study medications (bottles), numeric
- Medication names (bottle 1 med, bottle 2 med, bottle 3 med)
- 7.2 Baseline Medication Use Questionnaire:
  - 3-item questionnaire: Please perform a linear transformation of the following three variables to a scale of 100 and take the mean of the three for each patient, for those with baseline survey data:
    - missed\_doses: numerical value, 0-30. For each day missed, calculate the percentage of days taken out of 30 (e.g. missed\_doses=2  $\rightarrow$  28/30 = 93.33)
    - medication supposed:
      - 1=Never → 0
      - 2=Rarely → 20
      - 3=Sometimes → 40
      - 4=Usually → 60
      - 5=Almost Always → 80
      - 6=Always → 100
    - meds good job:
      - 1=Very Poor  $\rightarrow$  0
      - 2=Poor → 20
      - $3=Fair \rightarrow 40$

- 4=Good → 60
- 5=Very Good → 80
- 6=Excellent → 100
- Please generate a flag for missing any one of these fields (missed\_doses, medication\_supposed, meds\_good\_job)
- Automaticity score categories (automaticity): Present the scores for the 4 questions automaticity 1 end to automaticity 4 end.
  - 0=No
  - 1=Yes
- Routine related questionnaire
  - Score the following from 1 (Not at all) to 7 (Very much so): routine, same\_time, continue\_way, take\_same\_place, take\_right\_before, take\_water, take\_same\_cup, keep same place
- Perception related questionnaire
  - Score from 1 (Strongly Disagree) to 5 (Strongly Agree) the following: regular\_apts, tx\_plan\_difference, med\_help\_control, prescribed\_take\_daily, not\_taking\_effect, feel well stop, live long, control gout, gout better worse, actions effect

### 7.3 Baseline Gout Questionnaire

- o gout 1 (1 = Yes, 0 = No)
- $\circ$  gout 2 (1 = Yes, 0 = No)
- $\circ$  gout 3 (1 = Yes, 0 = No)
- gout\_4 (Score from 1 to 10)

### 8. Outcome variables and study follow-up:

### A) Primary Outcome (Average daily adherence):

For each patient, please measure the following outcomes beginning on the index date:

- a) Follow-up period for each patient
  - Some patients may not have a full 18 weeks of follow-up. This is based on the time between the index date (start\_date) and the end date (study\_date) or (withdraw\_date) whichever is earlier in REDCap. Please provide the number of days between the index date and the end date in REDCap.
- b) Calculate daily adherence during the follow-up period (adh\_daily), using the available time stamps from the 352 daily **Pillsy files** merged with the **REDCap file:** 
  - 1. Daily adherence values are calculated from Pillsy files, while date information should be taken from REDCap file.
  - 2. Medications are named using "Medication # QD/BID" (drugName). If name includes "QD", count as 1 expected daily dose; if name includes "BID", count as 2 expected daily doses.
  - **3.** Time stamps (eventTime) within 3 hours of each other (e.g. 9:00am and 11:59am) should be collapsed into one dose. There will likely be multiple time stamps for each opening, but they should be counted as one dose.
  - **4.** Time stamps between 12:00am and 3:00am should be counted as taken on the previous calendar date (i.e., the day before).

- **5.** Adherence is calculated as taking all expected doses of medications, with each medication weighted equally.
  - E.g., If a patient has 1 QD med and 2 BID meds, their calculation would be (1/3)(X/1) + (1/3)(X/2) + (1/3)(X/2) = 1
- **6.** Please provide the calculated daily adherence values for all the patients as a separate dataset containing the record\_id and the calculated daily adherence values.
- 7. Separately, please also provide the daily adherence for Allopurinol QD only. This variable will later be used for sensitivity analysis. The daily adherence will be recorded as a binary variable (1/0) (adh daily allopurinolgd)
  - E.g., if a patient takes 1 QD Allopurinol, their adherence for that day would be either 1 or 0.
- c) Using these daily calculations, generate the following adherence measure outcomes:
  - 1. Aggregate adherence (adh\_daily) into the mean daily adherence value for each patient (ranging from 0 to 1) for the 18 weeks from "start\_date" to the end of follow up (if date range is less than 18 weeks, calculate just for the respective date range) → label this as "adherence primary outcome"
  - 2. Repeat the aggregation of adherence for each patient omitting the first 7 days of data (i.e., index date -> index date+7)
  - **3.** Repeat the aggregation of adherence for each patient omitting the first 14 days of data (i.e., index date -> index date+14)
  - **4.** Repeat the aggregation of adherence for each patient, but censor patients in the adherence calculation at the time they have stopped using the electronic pill bottle for >30 days (defined as "adh\_daily"=0 for >30 consecutive days in Pillsy data)
    - Please generate a flag for the patient (1/0) and provide the date in which they were censored if this occurs (leave the date as missing if does not occur)
  - **5.** Repeat the aggregation of adherence for each patient for the **12 weeks** from "start date" to the "intervention\_date" (the intervention completion date) or "withdraw\_date", whichever is earlier.
  - **6.** Repeat the aggregation of adherence (adh\_daily\_allopurinolqd) for 18 weeks from "start\_date" to the end of follow up for Allopurinol QD label as "adh\_allopurinol".
- d) Use generalized linear models (proc genmod) to compare nonadaptive vs. control and adaptive vs. control; calculate unadjusted mean differences for these groups and adjusted mean differences (adjusted for age, sex, race/ethnicity). The link=identity and dist=normal). Recruitment type (PCP vs. rheumatology) also accounted for in the model.

## B) Uric acid level outcomes (Change in uric acid levels – Exploratory outcome)

- a) Using the **REDCap file**:
  - Please measure the difference between "ua\_end" (outcome) and "ua\_baseline" (baseline).
  - o Please provide the dates for both "ua\_date\_end" and "ua\_baseline\_date"
  - Please provide a flag if missing "ua end" (outcome)
- b) Use generalized linear models (proc genmod) to compare nonadaptive vs. control and

adaptive vs. control; calculate unadjusted mean differences for these groups and adjusted mean differences (adjusted for age, sex, race/ethnicity). The link=identity and dist=normal). Recruitment type (PCP vs. rheumatology) and baseline uric acid level also accounted for in the model.

## C) Self-Reported Outcomes:

- Automaticity scores (automaticity): automaticity\_1\_end to automaticity\_4\_end.
  - 0=No
  - 1=Yes
- Routine related questionnaire
  - Score the following from 1 to 7: routine\_end, same\_time\_end, continue\_way\_end, take\_same\_place\_end, take\_right\_before\_end, take\_water\_end, take\_same\_cup\_end, keep\_same\_place\_end
- Perception related questionnaire
  - Score from 1 (Strongly Disagree) to 5 (Strongly Agree) the following: regular\_apts\_end, tx\_plan\_difference\_end, med\_help\_control\_end, prescribed\_take\_daily\_end, not\_taking\_effect\_end, feel\_well\_stop\_end, live\_long\_end, control\_gout\_end, gout\_better\_worse\_end, actions\_effect\_end

# D) Feasibility Outcomes:

Score from 1 (Strongly agree) to 5 (Strongly disagree) the following: cue\_useful,
 cue text useful, reward text useful

#### **Requested Results:**

Table 1: Baseline characteristics

| | Usual Care | Non-adaptive | Adaptive |
|---|---|---|---|
| N, (%) | | - | |
| Age<br>(Mean, SD)<br>(Median, IQR) | | | |
| Female (N, %) | | | |
| Partnered/ Marital status Married Living with partner/ Domestic partnership Widowed Divorced/ Separated Never married/ Single | | | |

| | · |
|---|---|
| Race White Black or African American American Indian/ Alaska Native Asian Native Hawaiian or Other Pacific Islander Hispanic/Latinx | |
| Education level Less than high school diploma High school diploma Some college College degree Graduate degree | |
| Employment Employed Job seeking Not job seeking Retired Disabled | |
| Baseline Uric acid (mg/dL) | |
| Medication Use Baseline Automaticity score (Mean, SD) Routine Perception Recruitment method Rheumatology (N, %) | |
| PCP (N, %) | |
| Self-reported medications on a daily basis (Mean, SD) | |
| Self-reported medications on a weekly basis (Mean, SD) | |
| Number of prescribed study medications (N, %) 1 2 3 | |
| Baseline self-reported adherence (Mean, SD) | |
| Disease activity (Mean, SD) | |
| Number of Pillsy bottles used in the study | |

| 1<br>2+ | |
|-------------------------|-------------|
| Patients (adaptive arm) | intensified |

Table 2: Primary and Secondary Outcomes

| | Control<br>Mean<br>(SD) | Non-adaptive intervention Mean (SD) | Adaptive<br>intervention<br>Mean (SD) | Unadjusted absolute<br>difference | | Adjusted absolute<br>difference | |
|---|---|---|---|---|---|---|---|
| | | | | (Non-<br>adaptive<br>vs<br>Control) | (Adaptive<br>vs<br>Control) | (Non-<br>adaptive<br>vs Control) | (Adaptive<br>vs Control) |
| Primary<br>Outcome: | | | | , | | | |
| Adherence | | | | | | | |
| Secondary<br>Outcome: | | | | | | | |
| Change in uric acid levels | | | | | | | |
| Change in automaticity | | | | | | | |
| Change in perception | | | | | | | |
| Change in sense of routine | | | | | | | |